CLINICAL TRIAL: NCT01928121
Title: Effectiveness of an Interdisciplinary, Nurse-coordinated Atrial Fibrillation Expert Program for Primary Care Patients - A Clustered Randomized Controlled Trial
Brief Title: Effectiveness of an Interdisciplinary, Nurse-coordinated Atrial Fibrillation Expert Program for Primary Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Heidbuchel, Prof. Hein Heidbuchel, MD, PHD, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: not yet applicable
Record Dates: First submitted 2013-08-19; First posted 2013-08-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Atrial Fibrillation
Keywords: nurse; expert program; primary care; implementation; interdisciplinary; effectiveness; disease management system
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AF expert program (Experimental): Care provided by the interdisciplinary, nurse-coordinated AF expert program
  Interventions: Other: Care provided by AF expert program
- Usual care (No Intervention)

INTERVENTIONS:
Other: Care provided by AF expert program
  Arms: AF expert program

SUMMARY:
The purpose of this study is to assess the effectiveness of a newly developed interdisciplinary nurse-coordinated AF expert program for primary care patients. Therefore a prospective, pragmatic clustered randomized controlled trial will be performed in general practices.

ELIGIBILITY:
Inclusion Criteria:

* Every newly diagnosed AF patient.
* Every AF patient who is not seen by a cardiologist or electrophysiologist in the past 2 years before inclusion.
* AF must be confirmed on electrocardiogram.
* Capable of providing written informed consent.
* Dutch speaking and verbally testable, without cognitive impairment.

Exclusion Criteria:

* AF patients who once received an arrhythmologic consult about AF prior to the start of the study.
* AF patients who have a systematic follow-up at a cardiologist prior to the start of the study.
* Terminally ill AF patients
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
cardiovascular events | after 1 year
  Combined endpoint of cardiovascular hospitalizations, cardiovascular deaths and unplanned cardiovascular visits.
  * Cardiac death: Cardiac arrhythmic, Cardiac non-arrhythmic, Vascular non cardiac
  * Cardiovascular hospitalization: Arrhythmic events (AF, syncope, sustained ventricular tachycardia, cardiac arrest), Heart Failure, Acute myocardial infarction, Stroke, Systemic embolism, Major bleeding, Life-threatening effects of drugs
  * Unplanned cardiovascular visits

SECONDARY OUTCOMES:
Guideline adherence | after 1 year
  * Does the medical record report a formal CHA2DS2-VASc score, HAS-BLED bleeding risk score and EHRA score?
  * Does the medical record report an appropriate prescription of antithrombotic treatment.
  * Does the medical record report an appropriate application of rate and rhythm (not if asymptomatic, if contraindicated and not in patients with permanent AF)
  * Does the medical record report an appropriate upstream therapy? (For example in heart failure patients, is the heart failure treated)
Hospitalization days and clinic visits | after 1 year
  * Number of outpatient (internal or neurological) clinic visits per year
  * Number of emergency room visits per year due to AF
  * Number of hospitalization days due to AF
  * Number of hospitalization days for cardiovascular reasons
  * Number of hospitalization days on intensive care due to AF
Perceived health | After 1 year
  Perceived health will be measured by the EuroQol Five Dimensional Questionnaire (EQ-5D-3L)
AF related symptoms and symptom burden | After 1 year
  AF related symptoms and symptom burden will be measured by the Leuven Arrhythmia Questionnaire (LARQ)
Patient satisfaction | After year
  Patient satisfaction about information provided, about therapy and about follow-up, will be measured with a 10-point visual analog scale (VAS).
Patient knowledge | After 1 year
  The Atrial Fibrillation Knowledge Scale (AF knowledge scale) will be used.
Patient adherence with medication | After 1 year
  This will be assessed by self-report using the Dutch version of the 8-item Morisky Medication Adherence Scale (MMAS-8 scale).
Time to establishment of a management plan by electrophysiologist or cardiologist | After 1 year
  This outcome will be searched for by reviewing medical records of, or by interviewing, all participating patients at 1, 3, 6 months and 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium